CLINICAL TRIAL: NCT05222555
Title: A Phase 1b/2, Open-Label, Multicenter Study to Evaluate the Safety and Pharmacokinetics of a Modified Tafasitamab IV Dosing Regimen Combined With Lenalidomide in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Safety and Pharmacokinetics Study of a Modified Tafasitamab IV Dosing Regimen Combined With Lenalidomide in R-R DLBCL Patients
Acronym: MINDway
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR208C115; 2023-507993-42-00 (Registry Identifier: EU CT Number); 2021-003855-40 (EudraCT Number)
Record Dates: First submitted 2022-01-11; First posted 2022-02-03 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: monoclonal antibody; CD19; tafasitamab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Tafasitamab + Lenalidomide) (Experimental): Treatment:
  Tafasitamab will be combined with lenalidomide in R/R DLBCL patients.
  Dose:
  Cohort 1: The dose of tafasitamab will be level 1 high dose in combination with the approved dose
  Cohort 2: The dose of tafasitamab will be level 2 high dose in combination with the approved dose
  Expansion Cohort: The dose of tafasitamab will be the dose that is deemed safe and tolerable as determined from cohort 1 & cohort 2
  Treatment consisting of tafasitamab and lenalidomide combination will be administered until disease progression, unacceptable toxicity, or discontinuation for any other reason, whichever comes first. Lenalidomide can be given for up to 12 cycles in total, after which patients can continue with tafasitamab as monotherapy until progression or unacceptable toxicity.
  Interventions: Drug: Tafasitamab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Tafasitamab — tafasitamab will be administered intravenously at protocol defined timepoints
  Other Names: INCMOR00208; MOR00208; Xmab5574
Drug: Lenalidomide — lenalidomide will be administered orally at protocol defined timepoints

SUMMARY:
This is an open-label, multicentre study too Evaluate the Safety and Pharmacokinetics of a Modified Tafasitamab IV Dosing Regimen Combined with Lenalidomide (LEN) in Patients with Relapsed or Refractory Diffuse Large B-Cell Lymphoma (R/R DLBCL) who have had at least one, but no more than three prior systemic regimens and who are not eligible for high dose chemotherapy (HDC) with autologous stem-cell transplantation (ASCT) at the time of study entry.

ELIGIBILITY:
Major Inclusion Criteria:

1. Capable of giving signed informed consent
2. Age 18 years or older
3. Histologically confirmed diagnosis of DLBCL
4. Tumor tissue for retrospective central pathology review must be provided as an adjunct to participation in this study.
5. Patients must have:

   * relapsed and/or refractory disease
   * at least one bidimensionally measurable, PET positive disease site (transverse diameter of ≥1.5 cm and perpendicular diameter of ≥1.0 cm at baseline)
   * received at least one, but no more than three previous systemic regimens for the treatment of DLBCL and one therapy line must have included a CD20-targeted therapy
   * Eastern Cooperative Oncology Group 0 to 2
6. Patients not considered in the opinion of the investigator eligible to undergo intensive salvage therapy including ASCT
7. Patients must meet the following laboratory criteria at screening:

   * absolute neutrophil count ≥1.5 × 10^9/L
   * platelet count ≥90 × 10^9/L
   * total serum bilirubin ≤2.5 × ULN or ≤5 × ULN in cases of Glibert's Syndrome or liver involvement by lymphoma
   * alanine transaminase, aspartate aminotransferase and alkaline phosphatase ≤3 × ULN or <5 × ULN in cases of liver involvement
   * serum creatinine clearance ≥ 60 mL/minute
8. Patients who received previous CD19 targeted therapy (other than tafasitamab) must have CD19 positive lymphoma confirmed on a biopsy taken since completing the prior CD19 targeted therapy
9. Patients with primary refractory disease who received at least one, but no more than three previous systemic regimens (including a CD20 targeted therapy)

Major Exclusion Criteria:

1. Patients who are legally institutionalized or concurrent enrollment in another interventional clinical study
2. Patients who have:

   * other histological type of lymphoma
   * a history of "double/triple hit" genetics
3. Patients who have, within 14 days prior to Day 1 dosing:

   * not discontinued CD20-targeted therapy, chemotherapy, radiotherapy, investigational anticancer therapy or other lymphoma specific therapy
   * undergone major surgery (with 4 weeks) or suffered from significant traumatic injury
   * received live vaccines (within 4 weeks).
   * required parenteral antimicrobial therapy for active, intercurrent infections
4. Patients who:

   * have not recovered sufficiently from the adverse toxic effects of prior therapies
   * were previously treated with IMiDs® (e.g. thalidomide, LEN)
   * have history of hyper sensitivity to compounds of similar biological or chemical composition to tafasitamab IMiDs® and/or the excipients contained in the study treatment formulations
   * have undergone ASCT within the period ≤ 3 months prior to signing the informed consent form.
   * have undergone previous allogenic stem cell transplantation
   * have a history of deep venous thrombosis/embolism and who are not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period
   * concurrently use other anticancer or experimental treatments
5. History of other malignancy that could affect compliance with the protocol or interpretation of results. Exceptions

   * Patients with any malignancy appropriately treated with curative intent and the malignancy has been in remission without treatment for >2 years prior to enrollment are eligible
   * Patients with low-grade, early-stage prostate cancer (Gleason score 6 or below, Stage 1 or 2) with no requirement for therapy at any time prior to study are eligible
6. Patients with:

   * positive hepatitis B and/or C serology.
   * known seropositivity for or history of active viral infection with human immunodeficiency virus (HIV)
   * CNS lymphoma involvement
   * history or evidence of clinically significant cardiovascular, CNS and/or other systemic disease that would in the investigator's opinion preclude participation in the study or compromise the patient's ability to give informed consent
   * history or evidence of rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
   * gastrointestinal (GI) abnormalities (issue with absorption) including the inability to take oral medication
   * history or evidence of severe hepatic impairment (total serum bilirubin > 3mg/dL), jaundice unless secondary to Gilbert's syndrome or documented liver involvement by lymphoma
   * history of hypersensitivity to any of the study treatments or its excipients or to drugs of similar chemical class
   * any other medical condition which, in the investigator's opinion, makes the patient unsuitable for the study
7. Female participants: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods and refrain from breast feeding and donating eggs; agreement to ongoing pregnancy testing during the course of the study, and after study therapy has ended Male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom and agreement to refrain from donating sperm

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2027-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Director, Study Director — Incyte Corporation
Locations (62):
- United States (3):
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center - USOR, Dallas, Texas
  - Vista Oncology, Olympia, Washington
- Austria (3):
  - UK St. Pölten, Sankt Pölten, Lower Austria
  - Klinikum Wels Grieskirchen, Wels, Upper Austria
  - Universitatsklinikum Salzburg, Salzburg
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice V Praze, Prague
  - Fakultni nemocnice v Motole, Prague
- France (4):
  - Centre Hospitalier Universitaire Grenoble Alpes - Hopital Albert Michallon, Grenoble, Isère
  - CHU Nantes, Nantes, Loire-Atlantique
  - Centre Hospitalier Le Mans, Le Mans, Sarthe
  - CHU de Poitiers, Poitiers, Vienne
- Israel (5):
  - Soroka University Medical Centre, Beersheba, Southern District
  - Shamir Medical Center Assaf Harofeh, Be’er Ya‘aqov
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Medical Center - Hadassah Ein Kerem, Jerusalem
  - ZIV Medical Center, Safed
- Italy (8):
  - Ospedale Santa Maria Delle Croci, Ravenna, Emilia-Romagna
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Lombardy
  - ASST di Monza - Azienda Ospedaliera San Gerardo, Monza, Monza E Brianza
  - Fondazione del Piemonte per l'Oncologia (IRCCS), Candiolo, Piedmont
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliera di Perugia, Perugia, Umbria
- Poland (11):
  - Centrum Medyczne Poznan - PRATIA - PPDS, Skórzewo, Greater Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Dolnoslaskie Centrum Onkologii, Pulmonologii i Hematologii, Wroclaw, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Szpital Wojewodzki w Opolu, Opole, Opole Voivodeship
  - Szpitale Pomorskie Sp. z o. o., Gdynia
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - SPZOZ MiSWiA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Nasz Lekarz Osrodek Badan Klinicznych, Torun
- South Korea (12):
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggido
  - Dong-A University Medical Center, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Hanyang University Medical Center, Seoul
  - Asan Medical Center - PPDS, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (11):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Institut Catala d'Oncologia Girona, Girona
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital U. Infanta Leonor, Madrid
  - MD Anderson Madrid, Madrid
  - Hospital U. Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital U. Quironsalud Madrid, Madrid
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital U. Virgen del Rocio, Seville
  - Hospital Universitari La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Safety and Pharmacokinetics Study of a Modified Tafasitamab IV Dosing Regimen Combined With Lenalidomide in R-R DLBCL Patients — https://incyteclinicaltrials.com/studies/mor208c115

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 53 participants were enrolled at 26 study sites in Austria, Czech Republic, Israel, Italy, Poland, South Korea, Spain, and the United States through the data cutoff date of 17 July 2024.
Groups:
- Tafasitamab Dose Level 1 + 25 mg Lenalidomide: Tafasitamab was administered as an intravenous (IV) infusion in 28-day cycles until disease progression, unacceptable toxicity, or other criteria for treatment discontinuation were met. Lenalidomide 25 mg was administered once daily (QD) orally on Days 1 to 21 of each 28-day cycle for up to 12 cycles or until criteria for treatment discontinuation were met. Following discontinuation of lenalidomide, participants continued with tafasitamab monotherapy at the assigned treatment regimen.
- Tafasitamab Dose Level 2 + 25 mg Lenalidomide: Tafasitamab was administered as an IV infusion in 28-day cycles until disease progression, unacceptable toxicity, or other criteria for treatment discontinuation were met. Lenalidomide 25 mg was administered QD orally on Days 1 to 21 of each 28-day cycle for up to 12 cycles or until criteria for treatment discontinuation were met. Following discontinuation of lenalidomide, participants continued with tafasitamab monotherapy at the assigned treatment regimen.
Period: Overall Study
Arm/Group | Tafasitamab Dose Level 1 + 25 mg Lenalidomide | Tafasitamab Dose Level 2 + 25 mg Lenalidomide
Started | 6 | 47
Completed | 3 | 11
Not Completed | 3 | 36
Not completed — Ongoing | 2 | 18
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 6
Not completed — Withdrawal by Subject | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tafasitamab Dose Level 1 + 25 mg Lenalidomide | Tafasitamab Dose Level 2 + 25 mg Lenalidomide | Total
Number analyzed (Participants) | 6 | 47 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (10.49) | 71.9 (9.97) | 71.7 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 14 | 16
  Male | 4 | 33 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 44 | 49
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 18 | 18
  White | 6 | 27 | 33
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. Therefore, an AE could be any unfavorable or unintended sign (including an abnormal laboratory finding) or symptom temporally associated with the use of study treatment. A TEAE was defined as any AE that started or worsened after the first dose of study treatment until 90 days after the last dose of the study treatment. An AE that was present prior to study drug administration but increased in severity after treatment start was also included as a TEAE.
Time Frame: up to approximately 2 years
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug and had at least 1 postbaseline safety assessment. A valid safety assessment included death. Treatment groups were determined according to the actual treatment the participant received regardless of assigned study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafasitamab Dose Level 1 + 25 mg Lenalidomide | Tafasitamab Dose Level 2 + 25 mg Lenalidomide
Number analyzed (Participants) | 6 | 47
Participants | 6 | 45

2. Primary Outcome: Number of Participants With Any ≥Grade 3 TEAE
Description: The toxicity grade of TEAEs was graded using the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0) using the following definitions: Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: moderate; minimal; local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living (refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.). Grade 3: severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent intervention indicated. Grade 5: death related to AE.
Time Frame: up to approximately 2 years
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Tafasitamab Dose Level 1 + 25 mg Lenalidomide | Tafasitamab Dose Level 2 + 25 mg Lenalidomide
Number analyzed (Participants) | 6 | 47
Participants | 5 | 38

3. Secondary Outcome: Ctrough of Tafasitamab After 3 and 12 Treatment Cycles
Description: Ctrough was defined as the minimum concentration of tafasitamab.
Time Frame: predose on Cycle 3 Day 15; predose on Cycle 12 Day 28 (up to approximately 1 year [after twelve 28-day cycles])
Population: Pharmacokinetic Analysis Set: all participants who received at least 1 dose of tafasitamab and had at least 1 quantifiable serum tafasitamab concentration. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Tafasitamab Dose Level 1 + 25 mg Lenalidomide | Tafasitamab Dose Level 2 + 25 mg Lenalidomide
Number analyzed (Participants) | 6 | 28
micrograms per milliliter (μg/mL)
  Cycle 3 Day 15: number analyzed (Participants) | 4 | 28
  Cycle 3 Day 15 | 170 (117) | 228 (102)
  Cycle 12 Day 28: number analyzed (Participants) | 3 | 3
  Cycle 12 Day 28 | 87 (26) | 149 (69)

4. Secondary Outcome: Cmax of Tafasitamab After 3 Treatment Cycles
Description: Cmax was defined as the maximum observed plasma concentration of tafasitamab.
Time Frame: 30 minutes after the end of tafasitamab infusion on Cycle 3 Day 15 (up to approximately 85 days [after three 28-day cycles])
Population: Pharmacokinetic Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Tafasitamab Dose Level 1 + 25 mg Lenalidomide | Tafasitamab Dose Level 2 + 25 mg Lenalidomide
Number analyzed (Participants) | 4 | 28
micrograms per milliliter (μg/mL) | 792 (420) | 797 (273)

5. Secondary Outcome: Best Objective Response Rate (ORR) by Investigator Assessment up to Treatment Cycle 12
Description: ORR was defined as the percentage of participants with complete response (CR: disappearance of all evidence disease) or partial response (PR: regression of measurable disease and no new sites) as the best response achieved at any time during the study. Only responses of CR or PR that were documented before the initiation of new antilymphoma therapy (NALT) were considered. Response assessments were based on revised International Working Group response criteria for malignant lymphoma.
Time Frame: up to 19.8 months
Population: Full Analysis Set: all participants who received at least 1 dose of study treatment. Participants were analyzed according to the dose group to which they were initially assigned. Confidence intervals were calculated based on the Clopper-Pearson exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafasitamab Dose Level 1 + 25 mg Lenalidomide | Tafasitamab Dose Level 2 + 25 mg Lenalidomide
Number analyzed (Participants) | 6 | 47
percentage of participants | 50.0 [11.8 to 88.2] | 48.9 [34.1 to 63.9]

6. Secondary Outcome: Duration of Response (DoR) by Investigator Assessment
Time Frame: up to approximately 64 months (approximately 5 years)
Reporting Status: Not Posted, anticipated posting 2028-11

7. Secondary Outcome: Progression-free Survival (PFS) by Investigator Assessment
Time Frame: up to approximately 64 months (approximately 5 years)
Reporting Status: Not Posted, anticipated posting 2028-11

8. Secondary Outcome: Number of Participants Developing Anti-tafasitamab Antibodies up to Treatment Cycle 12
Description: Anti-tafasitamab antibody samples were defined as negative if they were screened or confirmed negative. Anti-tafasitamab antibody samples were defined as positive if they were positive in both the screening and the confirmatory assays.
Time Frame: up to approximately 1 year (after twelve 28-day cycles)
Population: Immunogenicity Analysis Set: all participants who received at least 1 dose of tafasitamab and had at least 1 valid anti-tafasitamab antibody assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Tafasitamab Dose Level 1 + 25 mg Lenalidomide | Tafasitamab Dose Level 2 + 25 mg Lenalidomide
Number analyzed (Participants) | 6 | 47
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to approximately 2 years
Description: Adverse events have been reported for the Safety Analysis Set, comprised of all participants who received at least 1 dose of study drug and had at least 1 postbaseline safety assessment. A valid safety assessment included death. Treatment groups were determined according to the actual treatment the participant received regardless of assigned study treatment.
Groups:
- Total: Total
Arm/Group | Tafasitamab Dose Level 1 + 25 mg Lenalidomide | Tafasitamab Dose Level 2 + 25 mg Lenalidomide | Total
All-Cause Mortality (participants affected / at risk) | 1/6 | 8/47 | 9/53
Serious Adverse Events (participants affected / at risk) | 2/6 | 20/47 | 22/53
Other Adverse Events (participants affected / at risk) | 6/6 | 40/47 | 46/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tafasitamab Dose Level 1 + 25 mg Lenalidomide (N=6) | Tafasitamab Dose Level 2 + 25 mg Lenalidomide (N=47) | Total (N=53)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 2 (3)
Asthenia (General disorders) | 0 (0) | 2 (2) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3) | 3 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tafasitamab Dose Level 1 + 25 mg Lenalidomide (N=6) | Tafasitamab Dose Level 2 + 25 mg Lenalidomide (N=47) | Total (N=53)
Alanine aminotransferase increased (Investigations) | 1 (2) | 2 (2) | 3 (4)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 9 (12) | 11 (16)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Asthenia (General disorders) | 1 (1) | 6 (7) | 7 (8)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Basal ganglia stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 4 (4) | 4 (4)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (5) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 7 (10) | 9 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (3) | 0 (0) | 1 (3)
Human polyomavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
Hypotension (Vascular disorders) | 1 (2) | 2 (3) | 3 (5)
Influenza like illness (General disorders) | 1 (2) | 0 (0) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 5 (5)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 6 (6) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 29 (45) | 31 (49)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (4) | 3 (4)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pityriasis rubra pilaris (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)
Procedural anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 8 (11) | 9 (12)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 10 (14) | 11 (15)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT05222555/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT05222555/SAP_001.pdf